CLINICAL TRIAL: NCT04099914
Title: Exploitation of a BAse of Genetic Data (Obtained by Next Generation SEquencing) for the Validation of a Clinical Algorithm for the Diagnosis of Recessive Cerebellar Ataxias
Brief Title: Validation of a Clinical Algorithm for the Diagnosis of Recessive Ataxias
Acronym: BASE-AAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Neurology Department, CHU de Strasbourg-France (Unknown); Genetic Department , CHU Montpellier-France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0431
Record Dates: First submitted 2019-09-09; First posted 2019-09-23 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Ataxia
Keywords: Cerebellar ataxia; Neurogenetics; Next generation sequence; Clinical algorithm
MeSH Terms: conditions — Ataxia; Cerebellar Ataxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Genetic database of approximately 150 patients with cerebellar ataxia, referred since September 2013 for exome analysis to the Montpellier University Hospital Center. The genetic data are from clinical exome capture sequencing with the Trusight One sequencing panel kit (www.illumina.com/trusightone), allowing exploration of approximately 5,000 human disease genes. Each sample is accompanied by a consent that allows genetic analysis and data processing. Each sample is also accompanied by clinical information, usually consisting of a clinical information sheet adapted to patients with genetic ataxias or clinical reports. These data are already accessible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The field of clinical diagnosis of recessive cerebellar ataxias (ARCA) is particularly complex and Next Generation Sequencing (NGS) techniques have revolutionized this neuro-genetic field. The current challenge is to optimize the analysis of genetic data generated by NGS because: the processing of data remains very laborious; diagnostic yeld less than 50%; the interpretation of the variants sometimes very difficult. For this purpose of optimization, the team of the University Hospital of Strasbourg has developed a computer algorithm based on 124 clinical and para-clinical parameters (derived from the data of the literature), useful to guide the genes to be targeted in priority by genetic analysis, in the context of a suspicion of ARCA (> 60 known genes); this algorithm was validated retrospectively in 834 patients with genetically confirmed ARCA (92% Sense, 95% Spec). However, these 834 patients are often the same as those described in the literature and used for the elaboration of the algorithm. This introduces a bias in the initial evaluation of the algorithm, which therefore requires validation in clinical practice, from a cohort of patients referred for suspected ARCA (with or without a found genetic mutation). At the same time, Montpellier's genetics laboratory has developed a bioinformatic method for the search for copy number variations (CNV) that can be applied in a targeted manner to the genes predicted by the algorithm.

The principal aim of this study is the validation of a semi-automated clinical algorithm for NGS molecular diagnosis of ARCA; the secondary objective is to evaluate if the application of this algorithm coupled with a targeted bioinformatic analysis can increase the diagnostic yield of the NGS analysis.

DETAILED DESCRIPTION:
Design: Retrospective study based on clinico-genetic data. Total research duration: 22 months Plan of the study : More than 150 patients referred for ARCA suspicion have been analyzed by NGS (Montpellier platform) since September 2013. The clinical data of these patients will be entered at the computer level into the algorithm to obtain the prediction of the gene involved (under the form of a probability for each of the genes known to ARCA). The investigators will compare this result with that obtained by standard NGS analysis. For patients without molecular diagnosis defined after standard NGS analysis, the investigators will take the 5 most probable genes selected on the basis of the algorithm in order to carry out an in-depth analysis of the variants found and a bioinformatic analysis by semi-automatic detection of CNVs. Main Evaluation Criterion: Concordance of the algorithm with standard NGS analysis for the genetic diagnosis of ARCA. Secondary evaluation criterion:% of patients for whom the prediction based on the algorithm suggested the correct diagnosis (subsequently confirmed after revision in the detail of the genetic data) while the standard genetic analysis was not not informative. Statistical Analysis: The investigators will perform a concordance analysis (Cohen's k) to validate the algorithm in clinical practice. For a given patient, there will be concordance if: i) one of the first 5 genes predicted with the highest probability by the algorithm is compatible with the mutation found after standard NGS or ii) if no gene is predicted by the algorithm (score <20) and no mutation found by NGS analysis.

ELIGIBILITY:
Inclusion criteria:

- having a predominant phenotype of pure or complex cerebellar ataxia of probable genetic origin (after exclusion of acquired, inflammatory, tumoral, infectious or toxic forms) - having started before the age of 50; - evoking a modality of recessive transmission (sporadic cases, brothers or sister affected, consanguinity of the parents) - in which dominant genetic forms due to CAG expansion (SCA1, SCA2, SCA3, SCA6, SCA7) and pre-mutation of the FMR1 gene (if onset after age 45)

Exclusion criteria:

- objecting to the computer processing of the data contained in the medical file.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adut Patients with suspicion of recessive cerebellar ataxia , with onset before the age of 50 and with negative molecular analisys for Friedreich ataxia and dominant spinocerebellar ataxias due to trinucleotide expansion. .
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Agreement between the prediction of the algorithm and the result of the standard NGS analysis | 1 day
  In order to validate in clinical practice a semi-automated clinical algorithm designed to guide the molecular diagnosis obtained by Next Generation Sequencing (NGS) in patients with suspected Autosomal Recessive Cerebellar Ataxia (ARCA), we will measure the agreement between the prediction of the algorithm and the result of the standard NGS analysis. For each patient the agreement is defined as: 1) one of the first 5 gene predicted with the highest probability by the algorithm is also the mutated gene found after the NGS analysis; 2) if no gene is predicted by the algorithm (= none of the gene has a prediction score > 20) and no mutation is found after NGS analyses.

SECONDARY OUTCOMES:
Percentage of patients for whom the prediction based on the algorithm suggested the right diagnosis, while the standard NGS analysis was not informative | 1 day
  The secondary objective is to evaluate whether the application of this algorithm, coupled with a targeted bioinformatic analysis, changes the diagnostic yield compared to a NGS analysis performed in a conventional manner. Therefore, the secondary outcome will be the percentage of patients for whom the prediction based on the algorithm suggested the corrected diagnosis (confirmed in a second time after the review of the genetic data derived from NGS after the application of a targeted bioinformatic analysis), while the standard NGS analysis (blinded to algorithm prediction) was not informative

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Marelli, MD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC